CLINICAL TRIAL: NCT03099629
Title: Efficacy of Inspiratory Muscle Training on Respiratory Performance in Patients With Esophageal Cancer Receiving Combined Modality Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yu-Jen Chen, VS. Division of Radiation Oncology, Department of Radiology, Mackay Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 13MMHIS300
Record Dates: First submitted 2017-03-14; First posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Esophageal Cancer
Keywords: Inspiratory muscle training; Diaphragmatic surface electromyography; Respiratory muscle strength; Functional capacity
MeSH Terms: conditions — Esophageal Neoplasms

ARMS (1):
- IMT (Experimental): inspiratory muscle training
  Interventions: Behavioral: inspiratory muscle training

INTERVENTIONS:
Behavioral: inspiratory muscle training — inspiratory muscle training will start with an intensity of 30% of maximal inspiratory pressure, 15 times/set, 3 sets/day, 7 days/week and training will continue until surgery is scheduled or 2 weeks after the completion of treatment if surgery is not suitable.

SUMMARY:
The purpose of this study is to investigate the effectiveness of inspiratory muscle training (IMT) on respiratory performance in patients with esophageal cancer during combined modality therapy.

DETAILED DESCRIPTION:
Background and Purpose: Incidence rates of esophageal cancer remain high in Eastern Asia. In 2012, esophageal cancer was the 9th leading cause of cancer deaths in Taiwan. Whether surgical resection is possible, combined modality therapy is usually required for the treatment of esophageal cancer. In clinical observation, patients underwent combined modality therapy usually demonstrated respiratory muscle dysfunction which might further impair physical activity and quality of life. The purpose of this study is to investigate the effectiveness of inspiratory muscle training (IMT) on respiratory performance in patients with esophageal cancer during combined modality therapy.

Methods: This is a prospective interventional study design. A total of 45 patients with newly diagnosed esophageal cancer will be recruited from the Mackay Memorial Hospital. All tests will be performed at baseline (prior to cancer treatment), weekly during treatment, prior to surgery, and one month after surgery. Tests will include demographic data collection, respiratory muscle performance (maximal inspiratory and expiratory pressure tests combined with diaphragmatic surface electromyography, and pulmonary functional test), dyspnea, and the functional exercise test (6-min walk test). IMT will start with an intensity of 30% of maximal inspiratory pressure, 15 times/set, 3 sets/day, 7 days/week and training will continue until surgery is scheduled or 2 weeks after the completion of treatment if surgery is not suitable. Repeated measure ANOVA will be used for analyzing difference of parameters among various time points.

Clinical relevance: The results of this study will help to better understand the clinical beneficial effects (e.g., better functional capacity) of an added inspiratory muscle training during combined modality therapy in patients with esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed primary esophageal cancer, aged more than 20 years, communicate without difficulty.

Exclusion Criteria:

* inability to perform inspiratory muscle training, the presence of unstable angina or myocardial infarction in recently one month, cannot cooperate with training protocols, and pregnancy.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Changes of maximal inspiratory pressure (MIP) | Baseline and weekly during CCRT treatment (for a total of 4-5 weeks)
  Change from baseline MIP at the end of each week's CCRT treatment
Changes of maximal expiratory pressure (MEP) | Baseline and weekly during CCRT treatment (for a total of 4-5 weeks)
  Change from baseline MEP at the end of each week's CCRT treatment
Changes of diaphragmatic surface electromyography (EMGdi) | Baseline and weekly during CCRT treatment (for a total of 4-5 weeks)
  Change from baseline EMGdi at the end of each week's CCRT treatment
Changes of forced expiratory volume in one second (FEV1) | Baseline and weekly during CCRT treatment (for a total of 4-5 weeks)
  Change from baseline FEV1 at the end of each week's CCRT treatment
Changes of forced vital capacity (FVC) | Baseline and weekly during CCRT treatment (for a total of 4-5 weeks)
  Change from baseline FVC at the end of each week's CCRT treatment

SECONDARY OUTCOMES:
Changes of functional exercise capacity using 6-minute walking distance | Baseline and weekly during CCRT treatment (for a total of 4-5 weeks)
  Change from baseline 6-minute walking distance at the end of each week's CCRT treatment
Changes of dyspnea using Modified Borg Dyspnea score | Baseline and weekly during CCRT treatment (for a total of 4-5 weeks)
  Change from baseline Modified Borg Dyspnea score at the end of each week's CCRT treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan